CLINICAL TRIAL: NCT04474938
Title: Efficacy of Daratumumab Combined With Bortezomib and Dexamethasone in Patients With Mayo 04 Stage III Light Chain Amyloidosis: a Prospective Phase II Clinical Trial
Brief Title: Daratumumab Combined With Bortezomib and Dexamethasone in Mayo 04 Stage III Light Chain Amyloidosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-AL2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Amyloidosis; Systemic
Keywords: light chain amyloidosis; daratumumab; bortezomib; hematologic response; prognosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dara-BD (Experimental): Daratumumab combined with bortezomib and dexamethasone
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — 16mg/kg, QW Cycles 1-2 (28 days/cycle), Q2W Cycles 3-6, and Q4W thereafter for up to 1 year
Drug: Bortezomib — 1.3mg/m2 of subcutaneous bortezomib on days 1, 8, 15 and 22 of a 28-day cycle for 6 cycles
Drug: Dexamethasone — 20mg of dexamethasone on days 1, 8, 15 and 22 of a 28-day cycle for 6 cycles

SUMMARY:
Patients with light chain (AL) amyloidosis who have advanced cardiac damage are at risk of premature mortality. There is ongoing unmet need for effective therapies to rapidly induce deep hematologic response and decrease the early death rate. Lately, trials of daratumumab in newly-diagnosed and relapsed/refractory AL amyloidosis have shown dramatic response rates. However, the benefits of upfront daratumumab in stage III AL patients, especially stage IIIb patients, have not yet been demonstrated definitely in prospective studies. Therefore, we designed a phase II, single arm clinical trial to investigate the efficacy and safety of co-administration of daratumumab with bortezomib and dexamethasone (BD) regimen in treatment-naïve patients with Mayo 04 stage III AL amyloidosis. We planned to enroll 40 patients, who would receive daratumumab and BD treatment for a total duration of 12 months. The primary endpoint is complete response and very good partial response at 3 months after treatment initiation. Secondary endpoints include overall survival, organ response and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old adults.

  * Biopsy proved treatment-naïve AL amyloidosis.
  * Mayo 2004 stage III.
  * dFLC > 50mg/L.
  * Patient must provide informed consent.

Exclusion Criteria:

* Co-morbidity of uncontrolled infection.
* Co-morbidity of other active malignancy.
* Co-diagnosis of multiple myeloma or waldenstrom macroglobulinemia.
* Co-morbidity of grade 2 or 3 atrioventricular block.
* Co-morbidity of sustained or recurrent nonsustained ventricular tachycardia.
* Seropositive for human immunodeficiency virus.
* Seropositive for hepatitis B (positive test for HBsAg). Participants with resolved infection (ie, HBsAg negative but positive for anti-HBc and/or anti-HBs) must be screened of HBV-DNA. Those who are PCR positive will be excluded.
* Seropositive for hepatitis C (except in the setting of a sustained virologic response).
* Grade 2 or higher neuropathy according to National Cancer Institute Common Terminology Criteria for Adverse Events.
* Neutrophil <1×10E9/L，hemoglobin < 7g/dL，or platelet < 75×10E9/L.
* Severely compromised hepatic or renal function: ALT or AST > 2.5 × ULN, total bilirubin > 1.5mg/dL，or eGFR < 40mL/min (those with renal dysfunction due to renal involvement or renal hypoperfusion from cardiac amyloidosis could be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Hematologic very good partial response or better at 3 months after treatment initiation | 3 months
  Very good partial response or better is defined as complete response or very good partial response. Complete response: normalization of free light chain levels and ratio with negative serum and urine immunofixation electrophoresis. Very good partial response: difference between involved and uninvolved free light chains (dFLC) less than 40 mg/L

SECONDARY OUTCOMES:
Overall survival | 2 years
major organ deterioration progression-free survival | 2 years
Time to next treatment | 2 years
Mortality within 1 month from treatment initiation | 1 month
Mortality within 3 months from treatment initiation | 3 months
Mortality within 6 months from treatment initiation | 6 months
Hematologic very good partial response or better at 1 month after treatment initiation | 1 month
Hematologic very good partial response or better at 6 months after treatment initiation | 6 months
Hematologic very good partial response or better at 12 months after treatment initiation | 12 months
Stringent dFLC response | 1 year
  dFLC declined to less than 10 mg/L
Time to hematologic response | 1 year
Organ response at 3 months after treatment initiation | 3 months
Organ response at 6 months after treatment initiation | 6 months
Organ response at 12 months after treatment initiation | 12 months
Time to cardiac response | 1 year
Time to liver response | 1 year
Time to renal response | 1 year
Adverse events | treatment initiation to 30 days after last dose of treatment
  Adverse events are collected until 30 days after last dose of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No